CLINICAL TRIAL: NCT05783752
Title: Effects of Stair Stepping on Late Day Postprandial Glycemia
Brief Title: Short, Simple, Exercise to Improve Circadian Dependent Postprandial Glycemic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HS-2023-0003
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Postprandial Glycemic Response; Postprandial Hyperglycemia; Postprandial Insulin
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stair-Stepping then Control (Experimental): Participants start with stair-stepping 15 minutes after meals on day 1 followed by no exercise on day 2. Sequence continues throughout the 10 days.
  Interventions: Behavioral: Stair Stepping; Behavioral: No exercise control
- Control then Stair-Stepping (Experimental): Participants start with no exercise on day 1 followed by stair-stepping 15 minutes after meals on day 2. Sequence continues throughout the 10 days.
  Interventions: Behavioral: Stair Stepping; Behavioral: No exercise control

INTERVENTIONS:
Behavioral: Stair Stepping — 1 minute of stair-stepping (30 seconds up, 30 seconds down) at a self-selected pace identified on day 0 starting 15 minutes after each meal
Behavioral: No exercise control — Participants avoid exercise within 1 hour of eating a meal

SUMMARY:
The goal of this clinical trial is to test whether one minute of stair stepping at a comfortable pace can reduce blood sugar after meals. The main objectives of the study are:

Compare continuously measured post-meal glucose after stair-stepping to control condition Compare continuously measured post-meal glucose after stair-stepping between meals Assess interaction between condition and meal to determine if the effect of stair-stepping on post-meal glucose depends on meal

Participants will be in the study for 10 days and will be asked to:

Wear a continuous glucose monitor over the course of the study Perform either one minute of comfortable pace stair stepping 15 min after each meal OR no exercise 1 hour after eating a meal on alternating days Perform a dietary recall every two days Perform no exercise within one hour after each meal on any day during the study Consume no calories within one hour after each meal during the study

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants giving written informed consent will undergo a screening to determine eligibility for study entry. At day 1, patients who meet the eligibility requirements will be randomly assigned to Arm 1(stair stepping day followed by no exercise day sequence) or Arm 2(no exercise day followed by stair stepping day sequence). At this time participants will also be familiarized with the continuous glucose (i.e., blood sugar) monitor they will wear for ten days, be instructed how to fill out a food log every day and determine a comfortable stair stepping pace. On day 10 participants will return to the lab for sensor removal and transmitter return.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years
* able to climb and descend stairs
* access to stairs

Exclusion Criteria:

* glycemic medications that vary in dosage
* dosage from meal to meal or day to day (eg insulin titrated to meal size or carbohydrate content)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Postprandial Blood Glucose | continuous measure from meal consumption up to 1 hour post meal
  mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No